CLINICAL TRIAL: NCT02677766
Title: Occupational Therapy in Complex Patients: a Pilot Study
Acronym: TO_EFFI15_14
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stefania Costi (Other)
Collaborators: Azienda USL Reggio Emilia - IRCCS (Other Government)
Responsible Party: Sponsor-Investigator, Stefania Costi, MSc in PT, University of Modena and Reggio Emilia
Organization: University of Modena and Reggio Emilia (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TO_EFFI15_14
Record Dates: First submitted 2016-01-29; First posted 2016-02-09 (Estimated); Results first posted 2019-09-09 (Actual); Last update posted 2019-09-09 (Actual); Status verified 2019-09

CONDITIONS: Complex Patients in Rehabilitation Phase
Keywords: Occupational Therapy; Complex patients; Randomized controlled trial; Occupational performance problem; Rehabilitation Complexity Scale
MeSH Terms: interventions — Occupational Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Intervention of Occupational therapy consists of implementing plans of action focused on the occupational needs chosen by patients through COPM
  Interventions: Other: occupational therapy
- usual care (Active Comparator): Usual care consists in rehabilitation treatment delivered by a multidisciplinary team
  Interventions: Other: Usual care

INTERVENTIONS:
Other: occupational therapy — an intervention phase in the period of hospitalization for rehabilitation in the hospital, aimed mainly at achieving objectives related to the area of self-care and, secondly, the objectives in the areas of productivity and leisure, identified at T0; plus an intervention in the post-discharge at the patient's home, aimed primarily at achieving objectives related to the areas of productivity and leisure time and, secondly, to possible targets in residues of self-care, identified in T0.
  Arms: Intervention
Other: Usual care — Usual care consists in rehabilitation treatment delivered by a multidisciplinary team
  Arms: usual care

SUMMARY:
To date, there are no studies that demonstrate that the intervention of Occupational Therapy (OT) in patients considered to be complex, regardless of diagnosis, could improve clinical and functional outcome for the patient. For this reason, the investigators propose one randomized controlled trial that will compare the group receiving the intervention of OT and the control group, to quantify the level of performance and satisfaction in the activities of interest of the patient, identified through the COPM. The hypothesis is that the benefit may be higher, as clinically relevant, in the group of complex patients treated with the proposed intervention of OT compared to those receiving the usual rehabilitation therapy.

DETAILED DESCRIPTION:
The investigators already implemented an observational pilot study, aimed at defining the characteristics and needs of the population in question and the OT intervention characteristics. These information will now be used to implement this randomized controlled trial, designed to demonstrate the effectiveness of the OT intervention on the basis of clinically relevant outcome measures.

This study will be set with exploratory purposes, with appropriate high number, which will allow the investigators to quantify the difference between the two groups in terms of performance scores derived from the COPM (COPM_p). From the results of this part it will then depend on the planning for the subsequent study with the correct sample size.

ELIGIBILITY:
Inclusion Criteria:

* complex inpatient

Exclusion Criteria:

* primary psychiatric disorders,
* language barriers,
* severe cognitive impairment
* communication disability

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Arcispedale Santa Maria Nuova, Reggio Emilia, RE, Italy

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Pellegrini M, Formisano D, Bucciarelli V, Schiavi M, Fugazzaro S, Costi S. Occupational Therapy in Complex Patients: A Pilot Randomized Controlled Trial. Occup Ther Int. 2018 Sep 3;2018:3081094. doi: 10.1155/2018/3081094. eCollection 2018. PMID 30250407
- Available data/document: Clinical Study Report: TOEFFI15_14 — https://www.ncbi.nlm.nih.gov/pubmed/30250407 — Titolo dello studio: Terapia occupazionale nei pazienti complessi : studio pilota. Codice protocollo TOEFFI15_14 Data di rilascio: 16/09/15

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention | Usual Care
Started | 20 | 20
Completed | 15 | 17
Not Completed | 5 | 3

BASELINE CHARACTERISTICS:
Population: Ethnicity not collected
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Usual Care | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 13 | 20
  >=65 years | 13 | 7 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.35 (14.67) | 62.75 (10.99) | 64 (26.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 12 | 11 | 23
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Follow-up of the Performance Score at the Canadian Occupational Performance Measure
Description: The Canadian Occupational Performance Measure is a valid, evidence-based outcome measure designed to capture a client's self-perception of performance in everyday living, over time.
  The score is between 1 and 10, where 1 indicates poor performance and low satisfaction, respectively, while 10 indicates very good performance and high satisfaction
Time Frame: T0 is the baseline at the patient ammission in the rehabilitation Ward; T2 is the follow-up at end of the intervention, 45 days ± 15 days from discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Intervention | Usual Care
Number analyzed (Participants) | 15 | 17
units on a scale | 7.28 (1.67) | 4.77 (1.89)

ADVERSE EVENTS:
Time Frame: to the end of the study, which means 45 days post hosèital discharge
Arm/Group | Intervention | Usual Care
All-Cause Mortality (participants affected / at risk) | 2/20 | 2/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention (N=20) | Usual Care (N=20)
referred to other wards for clinical reasons (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-03-19): https://cdn.clinicaltrials.gov/large-docs/66/NCT02677766/Prot_SAP_000.pdf